CLINICAL TRIAL: NCT01849770
Title: A Safety and Tolerability Study of Mexiletine in Patients With Sporadic Amyotrophic Lateral Sclerosis (SALS)
Brief Title: Mexiletine in Sporadic Amyotrophic Lateral Sclerosis (SALS)
Acronym: MX-ALS-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Michael D Weiss, Associate Professor, Department of Neurology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 43708
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Results first posted 2015-10-12 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Sporadic Amyotrophic Lateral Sclerosis
Keywords: SALS; Mexiletine; Safety
MeSH Terms: conditions — Amyotrophic lateral sclerosis 1 | interventions — Mexiletine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mexiletine, 300 milligrams (Active Comparator): Mexiletine, 300 milligrams by mouth per day for 12 weeks.
  Interventions: Drug: Mexiletine
- Mexiletine, 900 milligrams (Active Comparator): Mexiletine, 900 milligrams by mouth per day for 12 weeks.
  Interventions: Drug: Mexiletine
- Placebo (Placebo Comparator): Placebo, by mouth per day for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mexiletine
  Other Names: Mexitil
  Arms: Mexiletine, 300 milligrams; Mexiletine, 900 milligrams
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this research is to find out if mexiletine is safe and effective in people with Amyotrophic Lateral Sclerosis (ALS). In this trial, participants will be taking either 300 milligrams per day of mexiletine, 900 milligrams per day of mexiletine or placebo (non-active study drug). The safety and efficacy of these doses will be compared to see if one dose is better than the other.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a neurodegenerative disorder affecting primarily motor neurons, for which treatment designed to slow or arrest progression remains lacking. Mexiletine is a use-dependent sodium channel blocker that has been FDA-approved for decades for the treatment of cardiac arrhythmias and more recently to treat neuropathic pain in diabetic polyneuropathy. Mexiletine has been shown also to be protective of neurons following spinal cord, head injury, and cerebral ischemia, largely by blocking excitotoxicity. Based on previous studies, mexiletine appears to penetrate into the central nervous system at concentrations sufficient to confer significant protection. Recent unpublished studies in the laboratory of Dr. Robert Brown at the University of Massachusetts have also demonstrated that mexiletine ingestion in mice genetically engineered to express high levels of mutant cytosolic copper-zinc superoxide dismutase-1 (SOD1) transgene prolongs survival in these animals. As mexiletine already has FDA-approval as an anti-arrhythmic agent, much is known about the pharmacology and safety of this drug in non-ALS patients. We anticipate that by excluding subjects with a known history of cardiac disease and with the known neuroprotectant properties of this medication, mexiletine is a good choice for further study in an ALS clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Sporadic Amyotrophic Lateral Sclerosis (SALS) diagnosed as possible, laboratory-supported probable, probable, or definite ALS as defined by revised El Escorial criteria.
* Age 18 years or older.
* Disease duration ≤ 36 months from ALS symptom onset.
* Capable of providing informed consent and following trial procedures.
* Subjects must not have taken riluzole for at least 30 days or be on a 50 milligrams twice daily dose of riluzole for at least 60 days prior to randomization (riluzole-naïve subjects are permitted in the study).
* Subjects must not have taken medication for muscle cramping such as cyclobenzaprine, baclofen, carisoprodol, or methocarbamol, for at least 30 days prior to randomization or be on a stable dose for at least 60 days prior to randomization.
* Geographic accessibility to the site.
* Women must not become pregnant for the duration of the study and must be willing to use two contraceptive therapies and have a negative pregnancy test throughout the course of the study.
* Slow vital capacity (SVC) measure greater than or equal to 50% of predicted for gender, height, and age at the screening visit.
* Subjects medically able to undergo lumbar puncture (LP) as determined by the investigator (for example, no bleeding disorder, allergy to local anesthetics, a skin infection at or near the LP site, or evidence of high intracranial pressure).
* Must be able to swallow capsules throughout the course of the study, according to Principal Investigator (PI) judgment.
* Must have a caregiver assist with dispensing the study drug.

Exclusion Criteria:

* Invasive ventilator dependence, such as tracheostomy.
* Creatinine level greater than 1.5 milligram/deciliter.
* Serum glutamic oxaloacetic transaminase or (aspartate transaminase) / serum glutamic pyruvic transaminase (alanine aminotransferase) greater than 3 times the upper limit of normal at screening.
* History of known sensitivity or intolerability to mexiletine or lidocaine.
* Any history of either substance abuse within the past year, unstable psychiatric disease, cognitive impairment, or dementia.
* Clinically significant conduction abnormalities on electrocardiogram or a known history of cardiac arrhythmia.
* Known history of epilepsy.
* Known history of congestive heart failure (CHF) or history of myocardial infarction within the past 24 months.
* Use of mexiletine for 60 days prior to Baseline Visit.
* Exposure to any other experimental agent (off-label use or investigational) including high dose creatine (greater than 10 grams a day) within 30 days prior to Baseline Visit.
* Use of amiodarone, flecainide, duloxetine, tizanidine, or clozapine.
* Pregnant women or women currently breastfeeding.
* Placement of Diaphragm Pacing System (DPS) device less than 60 days prior to Baseline Visit.
* Planned DPS device implantation after Baseline Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Weiss, MD, Principal Investigator — University of Washington Medical School
Locations (10):
- United States (10):
  - UCLA, Neuromuscular Research Center, Los Angeles, California
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts (Worcester) Memorial Medical Center, Worcester, Massachusetts
  - Washington University Medical School, St Louis, Missouri
  - SUNY Upstate Medical Center, Syracuse, New York
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- See also: Northeast ALS Consortium Website — http://www.alsconsortium.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject in the study was enrolled July 23, 2013. Subjects were recruited and seen at Amyotrophic Lateral Sclerosis (ALS) clinics at 10 sites across the United States (U.S.).
Pre-assignment Details: Seventy-five (75) subjects signed the consent form and were considered enrolled in the study. Fifteen (15) subjects did not meet eligibility criteria and were considered screen failures. Sixty (60) subjects were randomized to one of three treatment arms. One (1) subject was randomized to the 900mg group but never started study drug.
Groups:
- Mexiletine, 300 Milligrams: Mexiletine, 300 milligrams by mouth per day for 12 weeks.
  Mexiletine
- Mexiletine, 900 Milligrams: Mexiletine, 900 milligrams by mouth per day for 12 weeks.
  Mexiletine
- Placebo: Placebo, by mouth per day for 12 weeks.
  Placebo
Period: Overall Study
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 900 Milligrams | Placebo
Started | 20 | 19 | 20
Completed | 20 | 15 | 19
Not Completed | 0 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 900 Milligrams | Placebo | Total
Number analyzed (Participants) | 20 | 19 | 20 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (7.1) | 58.0 (10.7) | 57.0 (7.0) | 58.0 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 10 | 23
  Male | 14 | 12 | 10 | 36
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 0 | 1
  Caucasian | 19 | 19 | 20 | 58
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 20 | 59
Months Since Symptom Onset [Mean (Standard Deviation); unit: Months] — Number of months since ALS symptom onset prior to enrolling into this study.
  Months | 21.0 (10.3) | 18.6 (9.2) | 17.5 (8.3) | 19.0 (9.3)
Months Since Diagnosis [Mean (Standard Deviation); unit: Months] — Number of months since enrolling into the study that a subject was diagnosed with ALS.
  Months | 8.6 (7.7) | 8.9 (8.2) | 7.3 (5.9) | 8.3 (7.2)
Slow Vital Capacity (Max % predicted) [Mean (Standard Deviation); unit: Max %-predicted] | 86.7 (19.1) | 86.2 (23.7) | 83.7 (22.6) | 85.6 (21.5)
Body Mass Index (BMI) (kg/m^2) [Mean (Standard Deviation); unit: kilograms (kg)/meter squared (m^2)] | 28.1 (5.1) | 27.3 (4.1) | 27.1 (3.3) | 27.5 (4.2)
Baseline Cramps in Previous 24 hours [Mean (Standard Deviation); unit: Number of Cramps] | 1.97 (3.06) | 1.68 (1.63) | 2.15 (2.13) | 1.94 (2.31)
Baseline Cramps in Previous 30 Days [Mean (Standard Deviation); unit: Number of Cramps] | 52.9 (91.0) | 29.1 (43.9) | 46.2 (55.9) | 42.8 (66.1)
Maximum Cramp Pain in Previous 24 hours [Mean (Standard Deviation); unit: units on a scale] — Cramp pain measured at 0 no pain and 10 is worst pain.
  units on a scale | 1.75 (2.24) | 2.32 (2.11) | 2.55 (2.78) | 2.20 (2.38)
Maximum Cramp Pain in Previous 30 Days [Mean (Standard Deviation); unit: units on a scale] — Cramp pain measured at 0 no pain and 10 is worst pain.
  units on a scale | 3.00 (2.38) | 3.37 (2.36) | 3.35 (2.70) | 3.24 (2.45)
ALSFRS-R Total Score [Mean (Standard Deviation); unit: units on a scale] — ALS Functional Rating Scale - Revised (ALSFRS-R) Total Score at Baseline. Scale is measured from 0 (worst score) to 48 points (best score).
  units on a scale | 36.3 (7.8) | 33.6 (6.7) | 34.9 (5.5) | 35.0 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Discontinued Study Drug
Description: Information on adverse effects of mexiletine will be determined at each visit by direct questioning of the subjects, clinical examination, review of concomitant medications, vital signs and laboratory test results.
Time Frame: Screening, Baseline Visit Pre-Dose and Post-Dose, Weeks 2, 6, and 12, and at the Final Safety Visit, if a subject discontinues study drug early. Adverse Events will be assessed via telephone Weeks 1, 10, and 16.
Measure: Number; unit: percentage of participants
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 900 Milligrams | Placebo
Number analyzed (Participants) | 20 | 19 | 20
percentage of participants | 5 | 32 | 5

2. Secondary Outcome: Trough Plasma Concentration (Cmin) of Mexiletine
Description: Subjects will have blood drawn to assess mexiletine concentrations for pharmacokinetics (PK) at the Week 6 Visit.
Time Frame: Week 6 Visit (pre-dose, hours 1, 2, 3, and 6 post-dose on Week 6)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 900 Milligrams | Placebo
Number analyzed (Participants) | 20 | 19 | 20
pg/mL | 0.23 (0.15) | 0.68 (0.38) | 0 (0)

3. Secondary Outcome: Peak Plasma Concentration (Cmax) of Mexiletine
Description: Subjects will have blood drawn to assess mexiletine concentrations for pharmacokinetics (PK) at the Week 6 Visit.
Time Frame: Week 6 Visit (pre-dose, hours 1, 2, 3, and 6 post-dose on Week 6)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 900 Milligrams | Placebo
Number analyzed (Participants) | 20 | 19 | 20
pg/mL | 0.41 (0.19) | 1.27 (0.67) | 0 (0)

4. Secondary Outcome: Area Under the Concentration Time Curve (AUC) of Mexiletine in Plasma.
Description: Subjects will have blood drawn to assess mexiletine concentrations for pharmacokinetics (PK) at the Week 6 Visit.
Time Frame: Week 6 Visit (up to 6 hours post dose)
Measure: Mean (Standard Deviation); unit: µg*hr/mL
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 900 Milligrams | Placebo
Number analyzed (Participants) | 20 | 19 | 20
µg*hr/mL | 2.34 (1.08) | 6.24 (3.18) | 0 (0)

5. Secondary Outcome: Mean Cerebrospinal Fluid (CSF)/Plasma Ratio
Description: The concentrations of Mexiletine were measured in cerebrospinal fluid (CSF) and plasma.
Time Frame: Week 6 Visit (up to 6 hours post dose)
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 900 Milligrams | Placebo
Number analyzed (Participants) | 20 | 19 | 20
ratio | 0.38 (0.15) | 0.46 (0.20) | 0 (0)

6. Secondary Outcome: Mean Weekly Cramp Frequency
Time Frame: Week 3-12, post titration of study medication
Measure: Mean (95% Confidence Interval); unit: cramps/week
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 900 Milligrams | Placebo
Number analyzed (Participants) | 20 | 19 | 20
cramps/week
  All Subjects n=20,19,20 | 0.785 [0.304 to 2.023] | 0.231 [0.125 to 1.250] | 2.505 [1.030 to 6.092]
  10+cramps previous 30 days at Baseline n=20,19,20 | 1.898 [0.494 to 7.288] | 0.595 [0.112 to 3.153] | 8.563 [3.217 to 22.79]

7. Other Pre Specified Outcome: Change in ALS Functional Rating Scale- Revised (ALSFRS-R) Score
Description: The ALSFRS-R is a quickly administered (5 minutes) ordinal rating scale (ratings 0-4) used to determine subjects' assessment of their capability and independence in 12 functional activities. All 12 activities are relevant in ALS. Initial validity was established by documenting that in ALS patients, change in ALSFRS-R scores correlated with change in strength over time, was closely associated with quality of life measures, and predicted survival.
Time Frame: Week 0, Week 2, Week 6, Week 12 (or Early Termination Date), and Week 16
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 900 Milligrams | Placebo
Number analyzed (Participants) | 20 | 19 | 20
scores on a scale
  Week 0 n=20,19,20 | 35.21 [32.9 to 37.5] | 35.21 [32.9 to 37.5] | 35.21 [32.9 to 37.5]
  Week 2 n=20,19,20 | 35.14 [32.7 to 37.6] | 34.58 [32.0 to 37.1] | 35.47 [33.0 to 37.9]
  Week 6 n=20,19,20 | 35.72 [33.1 to 38.3] | 33.08 [30.4 to 35.8] | 34.25 [31.7 to 36.8]
  Week 12 n=20,19,20 | 33.33 [30.4 to 36.3] | 31.85 [28.6 to 35.1] | 33.48 [30.5 to 36.4]
  Week 16 n=20,19,20 | 32.44 [29.2 to 35.7] | 31.94 [28.2 to 35.6] | 32.96 [29.7 to 36.2]
Statistical Analysis 1: Comparison: Mexiletine, 300 Milligrams vs Placebo; Test type: Superiority or Other; p = 0.561, Random slopes model; Slope = -0.23, 95% CI 2-sided [-1.03 to 0.56], Standard Error of Mean 0.40
Statistical Analysis 2: Comparison: Mexiletine, 900 Milligrams vs Placebo; Test type: Superiority or Other; p = 0.662, Random slopes model; Slope = -0.19, 95% CI 2-sided [-1.04 to 0.66], Standard Error of Mean 0.43

8. Other Pre Specified Outcome: Change in Slow Vital Capacity (SVC) Score
Description: The vital capacity (VC) (percent of predicted normal) will be determined, using the slow VC method. The SVC can be measured using conventional spirometers that have had a calibration check prior to subject testing. A printout from the spirometer of all SVC trials will be retained.
Time Frame: Week 0, Week 6, and Week 12 (or Early Termination Date)
Measure: Mean (95% Confidence Interval); unit: percent of predicted normal
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 900 Milligrams | Placebo
Number analyzed (Participants) | 20 | 19 | 20
percent of predicted normal
  Week 0 n=20,19,20 | 87.74 [80.0 to 95.5] | 87.74 [80.0 to 95.5] | 87.74 [80.0 to 95.5]
  Week 6 n=20,19,20 | 86.51 [78.1 to 94.9] | 82.92 [73.9 to 91.9] | 84.79 [76.3 to 93.3]
  Week 12 n=20,19,20 | 83.98 [75.1 to 92.8] | 77.18 [67.0 to 87.4] | 79.58 [70.7 to 88.4]
Statistical Analysis 1: Comparison: Mexiletine, 300 Milligrams vs Placebo; Test type: Superiority or Other; p = 0.178, Random slopes model; Slope = 1.71, 95% CI 2-sided [-0.80 to 4.22], Standard Error of Mean 1.25
Statistical Analysis 2: Comparison: Mexiletine, 900 Milligrams vs Placebo; Test type: Superiority or Other; p = 0.510, Random slopes model; Slope = -0.94, 95% CI 2-sided [-3.80 to 1.91], Standard Error of Mean 1.42

9. Secondary Outcome: Maximal Pain Severity
Description: At the Baseline Visit, subjects will be asked to recount the maximum intensity experienced with a muscle cramp in the previous 24 hours and the maximum intensity experienced with a muscle cramp in the previous 30 days.
  The visual analog scale (VAS) will be used to measures pain associated with muscle cramping. It will be used to measure muscle cramp intensity in this study. The scale rating is from 0-10; 0 equals no symptoms, 10 equals most severe symptoms.
  Subject will be provided with a muscle cramp diary to record muscle cramp intensity at home, daily.
Time Frame: Weeks 3-12, post titration of study medication
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 900 Milligrams | Placebo
Number analyzed (Participants) | 20 | 19 | 20
units on a scale
  All Subjects n=20,19,20 | 0.738 [0.364 to 1.494] | 0.340 [0.117 to 0.986] | 0.939 [0.466 to 1.893]
  10+cramps previous 30 days at Baseline n=20,19,20 | 1.348 [0.616 to 2.953] | 0.572 [0.176 to 1.859] | 2.033 [1.123 to 3.681]

10. Secondary Outcome: Cramp Frequency - Ratios for Comparisons of Doses for Weeks 3-12
Time Frame: Week 3-12, post titration of study medication
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | 300mg vs Placebo | 900mg vs Placebo
Number analyzed (Participants) | 20 | 19
ratio
  All Subjects n=20,19 | 0.313 [0.100 to 0.982] | 0.158 [0.050 to 0.495]
  10+cramps previous 30 days at Baseline n=20,19 | 0.222 [0.079 to 0.624] | 0.069 [0.013 to 0.374]

11. Secondary Outcome: Maximal Pain Severity - Ratios for Comparisons of Doses for Weeks 3-12
Time Frame: Week 3-12, post titration of study medication
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | 300mg vs Placebo | 900mg vs Placebo
Number analyzed (Participants) | 20 | 19
ratio
  All Subjects n=20,19 | 0.785 [0.342 to 1.802] | 0.361 [0.131 to 1.000]
  10+cramps previous 30 days at Baseline n=20,19 | 0.663 [0.347 to 1.267] | 0.281 [0.080 to 0.992]

12. Secondary Outcome: Mean Pain Severity
Description: as for outcome 9
Time Frame: Weeks 3-12, post titration of study medication
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 900 Milligrams | Placebo
Number analyzed (Participants) | 20 | 19 | 20
units on a scale
  All Subjects n=20,19,20 | 0.241 [0.115 to 0.509] | 0.136 [0.049 to 0.379] | 0.536 [0.275 to 1.046]
  10+cramps previous 30 days at Baseline n=20,19,20 | 0.467 [0.145 to 1.504] | 0.201 [0.050 to 0.812] | 1.248 [0.527 to 2.958]

13. Secondary Outcome: Mean Pain Severity - Ratios for Comparisons of Doses for Weeks 3-12
Time Frame: Week 3-12, post titration of study medication
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | 300mg vs Placebo | 900mg vs Placebo
Number analyzed (Participants) | 20 | 19
ratio
  All Subjects n=20,19 | 0.450 [0.183 to 1.110] | 0.254 [0.098 to 0.658]
  10+cramps previous 30 days at Baseline n=20,19 | 0.374 [0.135 to 1.035] | 0.161 [0.032 to 0.795]

ADVERSE EVENTS:
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 900 Milligrams | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/19 | 2/20
Other Adverse Events (participants affected / at risk) | 17/20 | 19/19 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mexiletine, 300 Milligrams (N=20) | Mexiletine, 900 Milligrams (N=19) | Placebo (N=20)
Balance Disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mexiletine, 300 Milligrams (N=20) | Mexiletine, 900 Milligrams (N=19) | Placebo (N=20)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 8 (15) | 2 (2)
Salivary Hypersecretion (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (6) | 0 (0)
Asthenia (General disorders) | 1 (1) | 3 (4) | 2 (2)
Chest Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Drug Withdrawal Syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (4) | 4 (7) | 3 (3)
Feeling Jittery (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gait Disturbance (General disorders) | 1 (2) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 1 (2) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ear Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Oral Herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 1 (2)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 5 (6) | 4 (7)
Joint Sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 2 (2) | 5 (5) | 2 (2)
Post Procedural Discomfort (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural Nausea (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 4 (5) | 2 (2)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Blood Glucose Increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood Potassium Decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood Pressure Diastolic Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Heart Rate Irregular (Investigations) | 0 (0) | 1 (1) | 0 (0)
Urine Analysis Abnormal (Investigations) | 1 (1) | 1 (1) | 0 (0)
Urine Output Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (3)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 (5) | 3 (3) | 3 (3)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Sensation of Heaviness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Balance Disorder (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Crying (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 6 (7) | 4 (4)
Dysarthria (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 4 (6) | 2 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Memory Impairment (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Muscle Contractions Involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 5 (7) | 1 (1)
Affect Lability (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (3) | 2 (2)
Euphoric Mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Heat Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Epidural Blood Patch (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0)
Surgical Stapling (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes